CLINICAL TRIAL: NCT01530308
Title: Early Pharmacological Intervention to Prevent Delirium: Haloperidol Prophylaxis in Older Emergency Department Patients
Brief Title: Haloperidol Prophylaxis in Older Emergency Department Patients
Acronym: HARPOON
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, Prabath W.B. Nanayakkara, Principal Investigator, Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NL38027.029.12; 2011-004762-15 (EudraCT Number); 3207 (Registry Identifier: Netherlands Trial Register (NTR))
Record Dates: First submitted 2011-12-22; First posted 2012-02-09 (Estimated); Last update posted 2015-11-26 (Estimated); Status verified 2015-11

CONDITIONS: Delirium
Keywords: Delirium
MeSH Terms: conditions — Delirium | interventions — Haloperidol; Antipsychotic Agents; Dopamine Antagonists; Butyrophenones

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Investigational medicinal product (Active Comparator): Haloperidol 1 mg twice daily at 12am and 20pm
  Interventions: Drug: Haloperidol
- Placebo group (Placebo Comparator): Placebo 1 mg twice daily at 12am and 20pm
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Haloperidol — An oral dosage of 1mg twice daily at 12am and 8pm.
  Other Names: Haldol; Antipsychotic agent; Dopamine antagonist; Butyrophenone
  Arms: Investigational medicinal product
Drug: Placebo — An oral dosage of 1mg twice-daily at 12am and 8 pm.
  Arms: Placebo group

SUMMARY:
The investigators propose a multicenter, randomized, double-blinded, placebo-controlled trial to study the effect of additive low-dose haloperidol prophylaxis on top of exciting care in a general population of older patients (age 70 years and over) acutely admitted to the hospital through the emergency department (ED) for general medicine and surgical specialties, and who are at-risk for developing in-hospital delirium on admission according to the VMS delirium risk questions (one or more positive answers out of three questions).

The investigators hypothesize that this intervention will reduce the incidence of in-hospital delirium as well as duration and severity of delirium.

DETAILED DESCRIPTION:
To address the aforementioned objectives, we propose a multicenter, randomized, double-blind, placebo-controlled clinical trial.

Eligible patients and/or their proxies will be verbally informed by the investigator on the content of the study, benefits and risks, and will receive a patient information folder on the nature of the study (version number, see appendix). The time to consider participation to the trial will be 4 hours maximum. Subsequently, the patient and/or their proxy will be asked for informed consent.

Subjects are screened for delirium-risk by the executive investigator administrating three delirium-risk questions to the patients or their care-givers, as recommended by the Dutch Safety Management (VMS) program:

1. Do you have memory complaints?
2. Did you need any help with activities of daily living in the past 24 hours?
3. During previous illness or hospital admission(s), did you have periods of confusion? One or more positive answers will identify at-risk patients. Eligible patients will be assigned a daily intervention with either low-dose haloperidol (an oral dosage of 1mg, twice-daily at 12pm and 8pm) or placebo by stratified randomization. The maximum intervention duration is 7 days. Hospital admission course of non at-risk patients according to the three VMS delirium-risk questions will be retrospectively assessed by medical chart review. Different study measurements will be collected on admission. A baseline ECG and standard ED laboratory will be done. Two additional blood samples of 10ml each will be drawn (one on admission and one at admission day 4) to determine haloperidol plasma levels and stored for future research. The investigator will assess baseline cognitive- and physical functioning on admission with different questionnaires and observational measures: the 6-item cognitive impairment test (CIT), the 6-item Index of Independence in Activities of Daily Living (ADL), the 8-item Instrumental Activities of Daily Living scale (IADL) and Informant Questionnaire on Cognitive Decline in the Elderly (IQCODE-N). The presence of delirium in the ED will be established according to the CAM-ICU and DSM-IV criterial. During admission, all subjects will receive the same 'high standard delirium care' based on effective non-pharmacological delirium intervention methods. Additionally to the standard ward rounds, the investigator will visit the patient at least on day 2, 4, and 8 for (extended) physical examination to evaluate any possible side-effects related to the intervention. According to protocol, an ECG is performed at least 24 hours (2 doses) and 72 hours (6 doses) after the first intervention dose, and if possible and the end of the study intervention period on request of the investigator. An ECG will be repeated at a 24-hour time-interval after every dose until a steady state is reached, when QTc >420ms-500ms on baseline ECG, or QTc prolongation >25% from baseline, of in case other QTc prolonging drugs are used. If QTc ≥ 500ms, the study medication will be discontinued. A list of QTC prolonging drugs contraindicated when using haloperidol (1st degree drug interactions, reason for action) is available and a warning system is implemented in the medication prescription system.

Development of delirium symptoms during the study will be evaluated by the Delirium Observation Screening (DOS) scale, administered 3 times per day. When delirium is suspected based on a mean DOS scale score >3/24 hours, the diagnosis is established according to the DSM-IV criteria by either the geriatrician or psychiatrist.

In case of established delirium within 7-day after initiation of the study intervention, administration of the assigned intervention is stopped since one of the primary endpoints (i.e. incidence) is reached. Unblinding will be performed immediately (24-hours a day, 7 days a week through the local hospital pharmacy at VUmc, procedures and argumentation will be recorded), and the treating physician will further decide on the treatment of the patients' delirium. Nursing staff will perform the DOS score 3-times daily to assess the duration of delirium, according to protocol. In addition, the investigator will assess delirium duration and severity with the DRS-R-98 once-daily. Both the DOS scale and DRS-R-98 are performed until delirium symptoms resolve or if participation in the study is no longer possible due to for example transfer to an other facility, ICU/CCU admission or death.

If no delirium symptoms develop within 7-days after initiation of the study intervention, administration of the assigned intervention treatment is stopped (after 14 doses). Further admission course will be evaluated by retrospective analysis of patients' charts. In patients discharged home within 7-days after initiation of the study intervention, study medication is aimed to be stopped the day before discharge since it takes approximately 12 - 38 hours to eliminate half of the originally administered oral haloperidol dose. These patients will be subjected to en extended physical examination on the day of discharge to evaluate any possible side-effects related to the intervention, if possible. The independent physician and researchers can be contacted for questions any time.

At the end of the study, all subjects' charts will be reviewed by one of the investigators.

During the follow-up period, an investigator will contact the subject and/or proxy by telephone, respectively at 3- and 6-months after hospital discharge, to evaluate physical function at that time with the ADL and IADL scale, and cognitive function with the 6-item CIT. Also, information on hospital re-admission(s), need for additional (health)care or (permanent) institutionalization after hospital discharge and death are reported. Each telephone conversation will take an estimated 20 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 70 years or over;
* The patient is at increased risk for developing in-hospital delirium on admission according to one or more positive answers on the VMS delirium-risk questions;
* The patient and/or proxy is able to provide written informed consent;
* The patient and/or proxy speaks either Dutch or English;
* The patient is admitted to the hospital for a general medicine or surgical specialty.

Exclusion Criteria:

* Patients presenting in the ED with delirium according to the DSM-IV criteria;
* Patients with clinically significant (cardiac) disorders: QTc interval prolongation (QTc ≥500ms), recent acute myocardial infarction, uncompensated heart failure (working diagnosis), acute coronary syndrome (ACS), arrhythmias treated with class IA and III antiarrhythmic medicinal products, history of ventricular arrhythmia, history of torsades, clinically significant bradycardia, second or third degree heart block, uncorrected hypokalaemia (potassium level 3.0 or lower);
* Patients with vascular dementia;
* Patients with Lewy Body dementia;
* Patients with Parkinson dementia;
* Patients with (a history of) hypokinetic movement disorders;
* Patients with (a history of) malignant neuroleptic syndrome;
* Patients with (a history of) serotonergic syndrome;
* Patients with (a history of) central anticholinergic syndrome;
* Patients who will be admitted to the oncology ward;
* Patients previously enrolled in the HARPOON study, or in other medical- or drug studies;
* Patients using QT prolonging drugs and/or medications of which concomitant use with haloperidol is contraindicated (clinically relevant drug interactions, 1st degree, listed in the appendix of the study protocol);
* Epilepsy;
* Substance abuse and dependence (DSM-IV criteria)
* Patients who are not able to take the study medication according to protocol (amendment)

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 242 (Actual)
Dates: Start 2012-11; Primary Completion 2015-04 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
The initial day and number of days there is a significant change from baseline in the mean Delirium Observation Screening (DOS) score, and/or delirium is diagnosed according to the DSM-IV criteria. | Assessed within 1 to 7 days after initiation of the study intervention.
  Reflecting the incidence, duration and severity of in-hospital delirium, which is the number of days in-hospital delirium is present in each participant who developed documented in-hospital delirium. Delirium symptoms are observed according to a mean Delirium Observation Screening (DOS) score >3 out of three DOS scale scores/24 hours (indicating significant change), and diagnosed according to meeting the DSM-IV delirium criteria.

SECONDARY OUTCOMES:
The number of days before there is a significant change from baseline in the mean Delirium Observation Screening (DOS) score, and delirium is diagnosed according to the DSM-IV delirium criteria. | Assessed from 1st day of inclusion, during the 7-day intervention period, up to delirium diagnosis or hospital discharge.
  Reflecting the time-to-develop delirium, which are the number of days from admission day until the first day delirium is diagnosed, assessed up to the day delirium develops during admission or participant is discharged from hospital. Delirium is diagnosed according to a mean Delirium Observation Screening (DOS) score >3 out of three DOS scale scores/24 hours (indicating significant change), and meeting DSM-IV criteria.
The (mean) number of days subjects are admitted to the hospital. | Assessed from 1st day of admission up to hospital discharge.
  The number of admission days per subject will be used to evaluate the mean hospital length of stay (LOS) in both study arms. The mean LOS is defined by the mean number of days each participant is admitted to hospital, assessed from admission day up to discharge date.
Functionality at baseline according to the Index of Independence in Activities of Daily Living (ADL) | 1 day of hospital admission.
  Functionality at baseline will be assessed according to the 6-item Index of Independence in Activities of Daily Living (ADL), administered on admission. Scores rang from 0-6 for both women and men, with higher scores indicating high function/independent.
Change from baseline functionality at 3 months according to the Index of Independence in Activities of Daily Living (ADL) | From baseline to assessment at time point 90 days after discharge date.
  Change from baseline functionality at 3 months after discharge date will be assessed at time point 90 days from hospital discharge date, according to the 6-item Index of Independence in Activities of Daily Living (ADL).
Change from baseline functionality at 6 months according to the Index of Independence in Activities of Daily Living (ADL). | From baseline to assessment at 180 days after discharge date.
  Change in functionality from baseline at 6 months after discharge date will be assessed at time point 180 days from hospital discharge date, according to the 6-item Index of Independence in Activities of Daily Living (ADL).
Functionality at baseline according to the Instrumental Activities of Daily Living Scale (IADL). | 1 day of hospital admission.
  Functionality at baseline will be assessed according to the 8-item Instrumental Activities of Daily Living Scale (IADL), administered on admission. Scores range from 0-8 for women, and 0-5 for men with higher scores indicating high function/independent.
Change from baseline functionality at 3 months according to the Instrumental Activities of Daily Living Scale (IADL). | From baseline to assessment at time point 90 days after discharge date.
  Change from baseline functionality at 3 months after discharge date will be assessed at time point 90 days from hospital discharge date, according to the 8-item Instrumental Activities of Daily Living Scale (IADL).
Change from baseline functionality at 6 months according to the Instrumental Activities of Daily Living Scale (IADL). | From baseline to assessment at time point 180 days after discharge date.
  Change in functionality from baseline at 6 months after discharge date will be assessed at time point 180 days from hospital discharge date, according to the 8-item Instrumental Activities of Daily Living Scale (IADL).
Mortality during hospital admission. | From 1st day of admission to the day that in-hospital death from any cause is documented admission, assessed up to hospital discharge.
  In-hospital mortality is reflected by the number of deaths (percentage of the total number of subjects included in the study) during hospital admission, assessed up to 30 days from admission date.
Overall mortality | From date of randomization until the date death from any cause is documented, assessed up to 180 days from hospital discharge date.
  Overall mortality is reflected by the number of deaths (percentage of the total number of subjects included in the study) from the date of randomization until the assessment time point at 180 days from admission date.

CONTACTS AND LOCATIONS:
Overall Officials: P WB Nanayakkara, Md, PhD, Principal Investigator — Amsterdam UMC, location VUmc; O J de Vries, MD, Principal Investigator — Amsterdam UMC, location VUmc; P M Bet, Pharm D, Principal Investigator — Amsterdam UMC, location VUmc
Locations (6):
- Netherlands (6):
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch, North Brabant
  - VUmc, Amsterdam, North Holland
  - Spaarne Ziekenhuis, Hoofddorp, North Holland
  - Medical Center Alkmaar, Alkmaar
  - Rijnland Ziekenhuis, Leiderdorp
  - Isala Klinieken, Zwolle

REFERENCES:
- [Derived] Schrijver EJ, de Vries OJ, Verburg A, de Graaf K, Bet PM, van de Ven PM, Kamper AM, Diepeveen SH, Anten S, Siegel A, Kuiperi E, Lagaay AM, van Marum RJ, van Strien AM, Boelaarts L, Pons D, Kramer MH, Nanayakkara PW. Efficacy and safety of haloperidol prophylaxis for delirium prevention in older medical and surgical at-risk patients acutely admitted to hospital through the emergency department: study protocol of a multicenter, randomised, double-blind, placebo-controlled clinical trial. BMC Geriatr. 2014 Aug 28;14:96. doi: 10.1186/1471-2318-14-96. PMID 25168927